CLINICAL TRIAL: NCT00769652
Title: The Influence of Changes in Body Composition on Quality of Life in Cancer Patients and The Impact of Medical Nutrition Therapy by a Registered Dietitian on Outcome
Brief Title: Medical Nutrition Therapy or Standard Care in Treating Patients With Lung Cancer, Pancreatic Cancer, or Stage III or Stage IV Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000592862; P30CA072720 (NIH); 000605 (Other: CINJ); 0220060217 (Other: UMDNJ IRB)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer; Malnutrition; Pancreatic Cancer; Prostate Cancer; Weight Changes
Keywords: malnutrition; non-small cell lung cancer; small cell lung cancer; stage III prostate cancer; stage IV prostate cancer; pancreatic cancer; weight changes
MeSH Terms: conditions — Lung Neoplasms; Malnutrition; Pancreatic Neoplasms; Prostatic Neoplasms; Body Weight Changes; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Nutrition Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical nutrition therapy (Experimental): Medical nutrition therapy
  Interventions: Behavioral: Medical nutrition therapy
- Standard care (Active Comparator): Standard care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Medical nutrition therapy — Medical nutrition therapy (MNT) refers to intervention with a registered dietitian or nutrition professional. MNT is a cyclical process which includes nutrition assessment, intervention, follow-up, and reassessment. Patients will receive a total of three (3) visits with the dietitian over a six-week period with follow-up during weeks 2-3 and weeks 6-9 based on their treatment schedule.
  Arms: Medical nutrition therapy
Behavioral: Standard Care — Standard nutritional care includes the National Cancer Institute's booklet "Eating Hints for cancer patients: before, during & after treatment".
  Arms: Standard care

SUMMARY:
This is a two-part study. Part I is an observational study. Part II is a randomized clinical trial to see how well medical nutrition therapy works compared with standard care in treating patients with lung cancer, pancreatic cancer, or stage III or stage IV prostate cancer.

DETAILED DESCRIPTION:
In Part II of the study, patients are stratified according to tumor type (pancreatic vs lung vs prostate). Patients are then randomized to 1 of 2 arms.

* Arm I (Medical nutrition therapy): intervention with a registered dietitian or nutrition professional. MNT is a cyclical process which includes nutrition assessment, intervention, follow-up, and reassessment. Patients will receive a total of three (3) visits with the dietitian over a six-week period with follow-up during weeks 2-3 and weeks 6-9 based on their treatment schedule.
* Arm II (standard care): Standard nutritional care includes the National Cancer Institute's booklet "Eating Hints for cancer patients: before, during & after treatment".

In both arms, patients' weight, fat free mass, and Patient Generated Subjective Global Assessment Score (PG-SGA) score will be assessed before, during, and after the intervention. The PG-SGA includes a patient report of symptoms and a healthcare professional assessment of medical, metabolic, and physical parameters.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with one of the following:

  * Pancreatic cancer
  * Lung cancer
  * Stage III or IV prostate cancer
* Undergoing treatment at The Cancer Institute of New Jersey

  * Are undergoing chemotherapy (part 2 only)
* Has lost ≥ 5% of their usual body weight in the previous 6 months (part 2 only)

PATIENT CHARACTERISTICS:

* Life expectancy > 60 days
* Must speak and read English
* Accessible in person or by phone for completing questionnaires
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Huhmann, DCN, RD, CSO, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight subjects were enrolled from October 2006 through May 2007 at Rutgers Cancer Institute of New Jersey, a comprehensive cancer center.
Pre-assignment Details: 1 subject was consented but did not get randomized.
Groups:
- Medical Nutrition Therapy: Medical nutrition therapy
  Medical nutrition therapy : Medical nutrition therapy (MNT) refers to intervention with a registered dietitian or nutrition professional. MNT is a cyclical process which includes nutrition assessment, intervention, follow-up, and reassessment. Patients will receive a total of three (3) visits with the dietitian over a six-week period with follow-up during weeks 2-3 and weeks 6-9 based on their treatment schedule.
- Standard Care: Standard care
  Standard Care : Standard nutritional care includes the National Cancer Institute's booklet "Eating Hints for cancer patients: before, during & after treatment".
Period: Overall Study
Arm/Group | Medical Nutrition Therapy | Standard Care
Started | 6 | 1
Completed | 6 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Nutrition Therapy | Standard Care | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (4.9) | 60 | 60.9 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Free Mass (FFM)
Time Frame: 3 years
Population: The study was closed early due to slow accrual and insufficient data was collected to analyze this outcome measure.
Arm/Group | Medical Nutrition Therapy | Standard Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Weight
Time Frame: 3 years
Population: The study was closed early due to slow accrual and insufficient data was collected to analyze this outcome measure.
Arm/Group | Medical Nutrition Therapy | Standard Care
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Patient Generated Subjective Global Assessment (PG-SGA) Score at Time of Initial Presentation and Throughout Study
Time Frame: 3 years
Population: The study was closed early due to slow accrual and insufficient data was collected to analyze this outcome measure.
Arm/Group | Medical Nutrition Therapy | Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Medical Nutrition Therapy | Standard Care
All-Cause Mortality (participants affected / at risk) | 5/6 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 0/6 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes